CLINICAL TRIAL: NCT02549261
Title: Nimotuzumab in Combination With Radiochemotherapy for Patients With Stage IIIA/IIIB Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-NI-LC-2
Record Dates: First submitted 2015-08-18; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: nimotuzumab; non-small cell lung cancer; radiochemotherapy; stage IIIA/IIIB non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- the tolerance trial of treatment (Experimental): nimotuzumab,chemotherapy (Cisplatin+Etoposide),radiotherapy,9 pts
  Interventions: Drug: nimotuzumab; Drug: Cisplatin; Drug: Etoposide; Radiation: radiotherapy
- A (Experimental): nimotuzumab,chemotherapy (Cisplatin+Etoposide),radiotherapy,9 pts
  Interventions: Drug: nimotuzumab; Drug: Cisplatin; Drug: Etoposide; Radiation: radiotherapy
- B (Placebo Comparator): chemotherapy (Cisplatin+Etoposide),radiotherapy,9 pts
  Interventions: Drug: Cisplatin; Drug: Etoposide; Radiation: radiotherapy

INTERVENTIONS:
Drug: nimotuzumab — the nimotuzumab treatment: 200mg/w weekly, for 16 weeks. A treatment:nimotuzumab for 3 levels (100mg/w, 200mg/w, 400mg/w, weekly, for 16 weeks).
  Arms: A; the tolerance trial of treatment
Drug: Cisplatin — Concurrent Chemotherapy,50mg/m2 (d1,d8),4 weeks/cycle, for 2 cycles. the consolidation chemotherapy: Cisplatin: 50mg/m2 (d1,d8)4 weeks/cycle, for 2 cycles.
Drug: Etoposide — Concurrent Chemotherapy, Cisplatin: Etoposide: 50mg/m2 (d1-5)，4 weeks/cycle, for 2 cycles.
  the consolidation chemotherapy:Etoposide: 50mg/m2 (d1-5)，4 weeks/cycle, for 2 cycles.
Radiation: radiotherapy — the tolerance trial of treatment A and B of treatment;95％PTV,60-66Gy/30-33/fraction,6-7weeks.

SUMMARY:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the efficacy and safety of the combination of Nimotuzumab administered concomitantly with chemoradiotherapy in patients with NSCLC .There is a tolerance trial of Nimotuzumab in Combination With Radiochemotherapy treatment before the randomization,double blind,muti-center sites trial of this treatment.

DETAILED DESCRIPTION:
There is a tolerance trial of Nimotuzumab in Combination With Radiochemotherapy treatment before the randomization,double blind,muti-center sites trial of this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70
2. both male and female
3. Subjects with pathologically or cytologically documented stage IIIB or IV NSCLC. Disease must be newly diagnosed.
4. Subjects would refer to the radical radiation therapy, but never have the previous chemotherapy or thoracic radiation therapy.
5. V20<30%, means that the percentage of the volume of lung which received the radiation<20Gy accounts the whole volume of lung is less than 30%.
6. Presence of at least 1 uni-dimensionally measurable index lesion,with the longest diameter ≥ 20 mm using conventional computer tomography(CT)/magnetic resonance imaging(MRI)scan or ≥ 10 mm using spiral computed tomography scan.
7. without pulmonary atelectasis, malignant pleural effusion malignant hydropericardium.
8. with ECOG performance status 0-2,and Life expectancy of more than 3 months.
9. without other malignancy history, except curative carcinoma in situ of cervix and skin basal cell carcinoma.
10. functions of major organs( haemogram,heart,liver,kidney)are basically normal, White blood count ≥3.5 x 109/L with neutrophils ≥1.5 x 109/L, platelet count≥100 x 109/L, and hemoglobin ≥90g/L.

    Total bilirubin ≤1.5 times upper limit of normal (ULN) range; alkaline phosphatase(ALP)≤ 2.5 times ULN, Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN, serum creatinine ≤ 1.2 times ULN .

    pulmonary function, FEV1≥1L, and >40% normal value.
11. willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
12. both female and male patients must use adequate methods of contraception.
13. Signature of the informed consent

Exclusion Criteria:

1. Previous radiotherapy, chemotherapy or anticancer biotherapy. Participation other clinical trials within 1 month prior to inclusion in the trial.
2. with the measureable lesion or lesion could be determined.
3. Severe diseases in lung, i.e. emphysema, interstitial pneumonia, bronchial asthma.
4. uncontrolled diabetes-random plasma glucose; RPG>11.1mmol/L.（RPG>11.1mmol/L, blood-fasting sugar; BFS; <7.8mmol/L，the patient also be enrolled）.
5. With other serious internal diseases or uncontrolled infection.
6. refractoriness dysentery or enterospasm, intestinal obstruction.
7. pregnancy, lactation, fertility but using a prohibited contraceptive method.
8. cardiovascular diseases history, congestive heart failure>GradeII, New York Heart Association (NYHA) criteria). With the unstable angina, de novo angina ( happened within 3 month prior to inclusion in the trial) or have myocardial in recently six months.
9. With drug addition, I.e. ,drug-taking, drug-taking for long time; type B hepatitis and C hepatitis in active stage, or with AIDS.
10. With organ transplantation,or using adrenocortical hormone or immunosuppressive agents for long time.
11. With history of serious allergic or allergy.
12. Not fit for the clinical trial judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12months

SECONDARY OUTCOMES:
Overall survival Time | 3 years
Quality of life | 12 months
Objective response rate | 12months
Disease controlled rate | 3 years
Adverse event rate | 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, profressor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China